CLINICAL TRIAL: NCT03806634
Title: Department of Physical Medicine & Rehabilitation, Taipei Veterans General Hospital
Brief Title: Development and Needs Assessment and Efficiency of Smart Communication System for Patients With ALS (Part 2)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-09-001A-2
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis, ALS, communication, needs
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research is aimed to asses the validity of the communication system improving the quality of life and the degree of sanctification of clinical patients and their caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Escorial revised criteria (Brooks et al., 2000),The diagnosis of ALS requires:

(A) the presence of:

* (A:1) evidence of lower motor neuron (LMN) degeneration by clinical, electrophysiological or neuropathologic examination (A:2) evidence of upper motor neuron (UMN) degeneration by clinical examination, and
* (A:3) progressive spread of symptoms or signs within a region or to other regions, as determined by history or examination, together with: (B) the absence of (B:1) electrophysiological or pathological evidence of other disease processes that might explain the signs of LMN and/or UMN degeneration, and (B:2) neuroimaging evidence of other disease processes that might explain the observed clinical and electrophysiological signs.

  * If they were Taiwanese and used traditional Chinese(Mandarin).
  * If they were older than age 20 years.

Exclusion Criteria:

* If they had been diagnosed with frontotemporal dementia, severe depression, or schizophrenia.
* If they cannot see the communication board after correction.
* If they cannot complete the questionnaire with researchers or family members help.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ALS were recruited from ALS clinics(Taipei Veterans General Hospital, Taiwan, R.O.C),20 participants. Participants were eligible for this study if they were diagnosed with definite, probable, probable laboratory-supported, or possible ALS according to the criteria (Brooks et al., 2000).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
System Usability Scale | 2019.04.01~2019.06.30
  It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. And also we can know the sanctification of the patient with ALS and their caregiver.

SECONDARY OUTCOMES:
Amyotrophic Lateral Sclerosis Specific Quality of Life Instrument-Revised, ALSSQOL-R | 2019.04.01~2019.06.30
  ALSSQOL-R is a 50 item instrument that measures overall quality of life (QOL) and six specific domains for individuals with ALS.
Taiwanese Depression Questionnaire, TDQ | 2019.04.01~2019.06.30
  The TDQ is a culturally relevant questionnaire, which is adaptable for screening depressive people in the local communities.
Caregiver Burden Scale | 2019.04.01~2019.06.30
  The burden experienced by family caregivers is the most important caregiver-related variable in care at home of a chronically-ill person. The extent of subjective burden has significant impact on the emotional and physical health of the family caregiver, and even influences the mortality of spouse caregivers. It affects the way the family caregiver deals with the care-receiver and determines the time of institutionalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, TW, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided